CLINICAL TRIAL: NCT06213870
Title: Screening of Endovascular Thrombectomy With MRI in Acute Ischemic Stroke
Status: Completed | Type: Observational
Sponsor: Tianjin Huanhu Hospital (Other)
Responsible Party: Principal Investigator, Ming Wei, Chief Physician, Tianjin Huanhu Hospital
Other Study IDs: TJHH-2023-WM51
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Fluid-attenuated Inversion Recovery Sequence Vascular Hyperintensity-diffusion-weighted Imaging Mismatch(FVH-DWI Mismatch); Image Evaluation; Endovascular Thrombectomy
Keywords: FVH-DWI mismatch;Endovascular Thrombectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MRI group: MRI Images were acquired on a 3T Siemens Prisma scanner (Siemens AG, Munich, Germany).Image sequences and typical parameter ranges were diffusion tensor imaging (repetition time [TR], 5200ms; echo time [TE], 80 ms; 4mm slice thickness; 40 slices) by using SE-EPI sequence; T1 imaging (TR, 240 ms; TE, 2.47 ms; 5 mm slice thickness; 17 slices) by using SE sequence;T2 imaging (TR, 4480 ms; TE, 99 ms; 4 mm slice thickness; 24 slices) by using FSE sequence; FLAIR imaging (TR, 8500 ms; TE, 95 ms; 5 mm slice thickness; 21 slices) by using IR sequence; time-of-flight magnetic resonance angiography images (TR, 20 ms; TE, 3 ms; 0.55 mm slice thickness; 40 slices) by using 3D-TOF sequence;
  In the MRI group, patients with FVH-DWI mismatch were considered to have EVT indications and were treated with EVT, while patients without FVH-DWI mismatch were treated with medication.
  Interventions: Diagnostic Test: Surgical criteria
- Perfusion group: The protocol of CT Perfusion was as follows: 100 mm coverage in the z-axis, tube voltage, 80 kV; tube current, 120 mA; section thickness, 5 mm. Twenty-four consecutive spiral acquisitions with 0.28 seconds of rotation time and 1.70 seconds of inter scan delay time were performed.
  Patients in the perfusion group were treated with EVT when there exist perfusion mismatch(defined as regional cerebral blood flow (<30%) was < 70 ml with mismatch ratio ≥ 1.8 and mismatch volume ≥ 15 ml), and were treated with medication when there was no perfusion mismatch.
  Interventions: Diagnostic Test: Surgical criteria

INTERVENTIONS:
Diagnostic Test: Surgical criteria — In the MRI group, patients with FVH-DWI mismatch underwent EVT surgery or were otherwise treated with medication.
  In the perfusion group, patients who meet the criteria of DEFUSE3 will receive EVT surgery, otherwise receive medication.

SUMMARY:
The goal of this observational study is to learn about the role of MRI evaluation based on FVH-DWI mismatch principle in preoperative evaluation of endovascular thrombolectomy.

The main questions it aims to answer are:

* The consistency between MRI and perfusion examination in determining EVT indications.
* The consistency of functional independence rate between patients screening with MRI and perfusion.

DETAILED DESCRIPTION:
MRI is the preferred imaging mode in many centers,for the diffusion-weighted imaging (DWI) sequences are highly sensitive to acute cerebral ischemia.In addition, MRI does not require intravenous contrast agent, which is simpler and more popular than perfusion.Fluid-attenuated inversion recovery (FLAIR)sequence vascular hyperintensity(FVH) is defined as focal, serpentine, or linear hyperintensity that usually occurs in the Sylvian fissure and is associated with large-vessel occlusion or stenosis.The FVH-DWI mismatch(defined as the FVH extended beyond the boundary of the DWI cortical lesions) had been confirmed has excellent sensitivity and specificity in predicting PWI-DWI mismatch.It is not well established whether MRI based on FVH-DWI mismatch and perfusion evaluation differ in determining EVT indications and outcomes.

The main objectives of this study were to (1) determine the proportion of patients eligible for EVT surgery selected by MRI based on FVH-DWI mismatch vs perfusion in a large multicenter registry and (2) identify statistical differences in functional outcomes and safety outcomes between the two evaluation methods.

Patients with ischemic stroke with anterior-circulation large-vessel occlusion in the late (6-24 h) time window from real-world, single center retrospective cohort registry were compared.In the MRI group, patients with FVH-DWI mismatch underwent EVT surgery or were otherwise treated with medication.In the perfusion group, surgical indications referring the DEFUSE 3 standards. The primary outcome was 90-day functional independence rate (mRS score ≤2) in all patients included(including EVT patient and medication patients).Safety outcomes included symptomatic intracranial hemorrhage (sICH), and 90-day mortality.

ELIGIBILITY:
Inclusion Criteria:

* (1) age ≥ 18 years old;
* (2) symptoms consistent with acute ischemic stroke and an onset time of 6-24h;
* (3) CT ASPECTS score≥6 points;NIHSS≥6points; modified Rankin scale (mRS) of 0-2 points prior to stroke;
* (4) internal carotid artery (ICA) and/or M1 segment of middle cerebral artery (MCA-M1) and M2 proximal segment occlusion with definite diagnosis.
* (5)agree to comply with the protocol follow-up requirements.

Exclusion Criteria:

* (1)Image unanalyzable.
* (2)3 months follow-up was not completed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were recruited in Tianjin Huanhu hospital in China between August 1, 2022, and Augut 1, 2023.
Sampling Method: Non-Probability Sample
Enrollment: 309 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
90-day functional independence rate | 90days
  Proportion of patients with mRS0-2 scores at 90 days

SECONDARY OUTCOMES:
symptomatic intracranial hemorrhage | 90days
  according to the definition proposed by European Cooperative Acute Stroke Study III: intracranial hemorrhage that is associated with deterioration in NIHSS of 4 or more points and the main reason for neurological deterioration

OTHER OUTCOMES:
90-day mortality | 90days
  Death from any cause within 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Ming Wei, PhD, Principal Investigator — Tianjin Huanhu Hospital
Locations (1):
- Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided